CLINICAL TRIAL: NCT02075151
Title: Bronchial Thermoplasty: Mechanism of Action and Defining Asthma Phenotype
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSRB/2013/00144
Record Dates: First submitted 2014-02-13; First posted 2014-03-03 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2014-02

CONDITIONS: Asthma
Keywords: Bronchial Thermoplasty
MeSH Terms: conditions — Asthma | interventions — Bronchial Thermoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bronchial Thermoplasty (Other): Bronchial thermoplasty
  Interventions: Procedure: Bronchial Thermoplasty

INTERVENTIONS:
Procedure: Bronchial Thermoplasty — Bronchial thermoplasty

SUMMARY:
According to World Health Organization (WHO) estimates, more than 200 million people suffer from asthma worldwide and in 2009, the disease had claimed 250,000 lives globally. Autopsy reports suggest 2 phenotypes of severe asthma: one that is characterized by intense airway inflammation with mucus plugging, and the other by severe bronchoconstriction causing respiratory failure in the absence of significant airway inflammation. However, it is not easy to stratify patients according to phenotypes without bronchoscopy. Although severe asthma comprises only 10% of affected individuals, it accounts for more than half of the total healthcare spending on asthma. Inhaled corticosteroids are effective by suppressing production of multiple pro-inflammatory mediators, unfortunately efficacy plateaus. Addition of long acting beta agonist and anti-cholinergic agent to inhaled corticosteroids offers some measure of relief but effective treatment of severe asthma remains an unmet goal, resulting in intensive utilization of healthcare resources. In 2010, the United States Food and Drug Administration (FDA) approved bronchial thermoplasty (BT) as an adjunctive therapy for severe asthma. BT is radiofrequency ablation of airway smooth muscle via bronchoscopy with each patient undergoing three procedures which targets different lobes of the lung 3 weeks apart. Studies have demonstrated improved symptom control allowing discontinuation of oral steroids in some patients as well as reductions in exacerbations, hospitalizations and use of rescue medications. No development of airway strictures or bronchiectasis, and regeneration of normal epithelium after BT has been observed. At present, it remains unclear if BT benefits all asthma phenotypes or if BT has any effect on airway inflammation and remodeling.

The hypothesis of this study is that bronchial thermoplasty is likely to benefit all severe asthma phenotypes, and achieves this by exerting an effect on airway inflammation and remodelling.

The specific aims of the study are: 1) to better define the asthma phenotype who will benefit from BT by microarray and gene expression profiling; 2) to study effects of BT on airway inflammation; 3) to define its role in the overall asthma management algorithm

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 21-65 years of age
* Poorly controlled severe persistent asthma (ACT score < 20) despite high-dose inhaled steroids (>500 mcg fluticasone/day or >800 mcg budesonide/day) in combination with inhaled long-acting Beta-2 agonist and/or anticholinergic agent. Other drugs include leukotriene modifiers, omalizumab (if used for at least 1 year prior), and oral corticosteroids 10mg/day or less
* Stopped smoking for > 1 year and <10 pack-years
* Stable maintenance asthma medications for 4 weeks
* Pre-bronchodilator FEV1 >60% predicted

Exclusion Criteria:

* Males and females <21 and >65 years of age
* Presence of pacemaker, internal defibrillator, or other implantable electronic devices
* Known sensitivity to medications required to perform bronchoscopy, including lignocaine and benzodiazepines
* Patients previously treated with Bronchial Thermoplasty (BT)
* Use of immunosuppressant (excluding oral steroids)
* Increased risk of adverse events associated with bronchoscopy or anesthesia (including pregnancy, uncontrolled coronary artery disease, acute or chronic renal failure, and uncontrolled hypertension)
* Inability to cease antiplatelet or anticoagulant therapy prior to procedure

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-02; Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Asthma Control Test (ACT) score | Up to 2 years

SECONDARY OUTCOMES:
Percentage of symptom-free days | Up to 2 years
Number of adverse events | Up to 2 years
Peak Expiratory Flow (PEF) | Up to 2 years
Exhaled nitric oxide (NO) | Up to 2 years
Forced Expiratory Volume in 1 Second (FEV1) | Up to 2 years
Non-contrast Computed Tomography (CT) scan of the thorax | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kay Leong Khoo, MD, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] HOUSTON JC, DE NAVASQUEZ S, TROUNCE JR. A clinical and pathological study of fatal cases of status asthmaticus. Thorax. 1953 Sep;8(3):207-13. doi: 10.1136/thx.8.3.207. No abstract available. PMID 13102418
- [Background] Kuyper LM, Pare PD, Hogg JC, Lambert RK, Ionescu D, Woods R, Bai TR. Characterization of airway plugging in fatal asthma. Am J Med. 2003 Jul;115(1):6-11. doi: 10.1016/s0002-9343(03)00241-9. PMID 12867228
- [Background] Saetta M, Di Stefano A, Rosina C, Thiene G, Fabbri LM. Quantitative structural analysis of peripheral airways and arteries in sudden fatal asthma. Am Rev Respir Dis. 1991 Jan;143(1):138-43. doi: 10.1164/ajrccm/143.1.138. PMID 1986670
- [Background] Hogg JC. Varieties of airway narrowing in severe and fatal asthma. J Allergy Clin Immunol. 1987 Sep;80(3 Pt 2):417-9. doi: 10.1016/0091-6749(87)90065-0. No abstract available. PMID 3624696
- [Background] Sur S, Crotty TB, Kephart GM, Hyma BA, Colby TV, Reed CE, Hunt LW, Gleich GJ. Sudden-onset fatal asthma. A distinct entity with few eosinophils and relatively more neutrophils in the airway submucosa? Am Rev Respir Dis. 1993 Sep;148(3):713-9. doi: 10.1164/ajrccm/148.3.713. PMID 8368644
- [Background] Good JT Jr, Kolakowski CA, Groshong SD, Murphy JR, Martin RJ. Refractory asthma: importance of bronchoscopy to identify phenotypes and direct therapy. Chest. 2012 Mar;141(3):599-606. doi: 10.1378/chest.11-0741. Epub 2011 Aug 11. PMID 21835905
- [Background] Haldar P, Pavord ID, Shaw DE, Berry MA, Thomas M, Brightling CE, Wardlaw AJ, Green RH. Cluster analysis and clinical asthma phenotypes. Am J Respir Crit Care Med. 2008 Aug 1;178(3):218-224. doi: 10.1164/rccm.200711-1754OC. Epub 2008 May 14. PMID 18480428
- [Background] Wahidi MM, Kraft M. Bronchial thermoplasty for severe asthma. Am J Respir Crit Care Med. 2012 Apr 1;185(7):709-14. doi: 10.1164/rccm.201105-0883CI. Epub 2011 Nov 10. PMID 22077066
- [Background] Lee P, Khoo KL. A review of current bronchoscopic interventions for obstructive airway diseases. Ther Adv Respir Dis. 2012 Oct;6(5):297-307. doi: 10.1177/1753465812455448. Epub 2012 Aug 9. PMID 22878625
- [Background] Venter JC, Adams MD, Myers EW, Li PW, Mural RJ, Sutton GG, Smith HO, Yandell M, Evans CA, Holt RA, Gocayne JD, Amanatides P, Ballew RM, Huson DH, Wortman JR, Zhang Q, Kodira CD, Zheng XH, Chen L, Skupski M, Subramanian G, Thomas PD, Zhang J, Gabor Miklos GL, Nelson C, Broder S, Clark AG, Nadeau J, McKusick VA, Zinder N, Levine AJ, Roberts RJ, Simon M, Slayman C, Hunkapiller M, Bolanos R, Delcher A, Dew I, Fasulo D, Flanigan M, Florea L, Halpern A, Hannenhalli S, Kravitz S, Levy S, Mobarry C, Reinert K, Remington K, Abu-Threideh J, Beasley E, Biddick K, Bonazzi V, Brandon R, Cargill M, Chandramouliswaran I, Charlab R, Chaturvedi K, Deng Z, Di Francesco V, Dunn P, Eilbeck K, Evangelista C, Gabrielian AE, Gan W, Ge W, Gong F, Gu Z, Guan P, Heiman TJ, Higgins ME, Ji RR, Ke Z, Ketchum KA, Lai Z, Lei Y, Li Z, Li J, Liang Y, Lin X, Lu F, Merkulov GV, Milshina N, Moore HM, Naik AK, Narayan VA, Neelam B, Nusskern D, Rusch DB, Salzberg S, Shao W, Shue B, Sun J, Wang Z, Wang A, Wang X, Wang J, Wei M, Wides R, Xiao C, Yan C, Yao A, Ye J, Zhan M, Zhang W, Zhang H, Zhao Q, Zheng L, Zhong F, Zhong W, Zhu S, Zhao S, Gilbert D, Baumhueter S, Spier G, Carter C, Cravchik A, Woodage T, Ali F, An H, Awe A, Baldwin D, Baden H, Barnstead M, Barrow I, Beeson K, Busam D, Carver A, Center A, Cheng ML, Curry L, Danaher S, Davenport L, Desilets R, Dietz S, Dodson K, Doup L, Ferriera S, Garg N, Gluecksmann A, Hart B, Haynes J, Haynes C, Heiner C, Hladun S, Hostin D, Houck J, Howland T, Ibegwam C, Johnson J, Kalush F, Kline L, Koduru S, Love A, Mann F, May D, McCawley S, McIntosh T, McMullen I, Moy M, Moy L, Murphy B, Nelson K, Pfannkoch C, Pratts E, Puri V, Qureshi H, Reardon M, Rodriguez R, Rogers YH, Romblad D, Ruhfel B, Scott R, Sitter C, Smallwood M, Stewart E, Strong R, Suh E, Thomas R, Tint NN, Tse S, Vech C, Wang G, Wetter J, Williams S, Williams M, Windsor S, Winn-Deen E, Wolfe K, Zaveri J, Zaveri K, Abril JF, Guigo R, Campbell MJ, Sjolander KV, Karlak B, Kejariwal A, Mi H, Lazareva B, Hatton T, Narechania A, Diemer K, Muruganujan A, Guo N, Sato S, Bafna V, Istrail S, Lippert R, Schwartz R, Walenz B, Yooseph S, Allen D, Basu A, Baxendale J, Blick L, Caminha M, Carnes-Stine J, Caulk P, Chiang YH, Coyne M, Dahlke C, Deslattes Mays A, Dombroski M, Donnelly M, Ely D, Esparham S, Fosler C, Gire H, Glanowski S, Glasser K, Glodek A, Gorokhov M, Graham K, Gropman B, Harris M, Heil J, Henderson S, Hoover J, Jennings D, Jordan C, Jordan J, Kasha J, Kagan L, Kraft C, Levitsky A, Lewis M, Liu X, Lopez J, Ma D, Majoros W, McDaniel J, Murphy S, Newman M, Nguyen T, Nguyen N, Nodell M, Pan S, Peck J, Peterson M, Rowe W, Sanders R, Scott J, Simpson M, Smith T, Sprague A, Stockwell T, Turner R, Venter E, Wang M, Wen M, Wu D, Wu M, Xia A, Zandieh A, Zhu X. The sequence of the human genome. Science. 2001 Feb 16;291(5507):1304-51. doi: 10.1126/science.1058040. PMID 11181995
- [Background] Verrills NM, Irwin JA, He XY, Wood LG, Powell H, Simpson JL, McDonald VM, Sim A, Gibson PG. Identification of novel diagnostic biomarkers for asthma and chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2011 Jun 15;183(12):1633-43. doi: 10.1164/rccm.201010-1623OC. Epub 2011 Mar 18. PMID 21471098
- [Background] Mann M, Hendrickson RC, Pandey A. Analysis of proteins and proteomes by mass spectrometry. Annu Rev Biochem. 2001;70:437-73. doi: 10.1146/annurev.biochem.70.1.437. PMID 11395414
- [Background] Naaby-Hansen S, Waterfield MD, Cramer R. Proteomics--post-genomic cartography to understand gene function. Trends Pharmacol Sci. 2001 Jul;22(7):376-84. doi: 10.1016/s0165-6147(00)01663-1. PMID 11431033
- [Background] Zhao J, Zhu H, Wong CH, Leung KY, Wong WS. Increased lungkine and chitinase levels in allergic airway inflammation: a proteomics approach. Proteomics. 2005 Jul;5(11):2799-807. doi: 10.1002/pmic.200401169. PMID 15996009
- [Background] Wong WS, Zhao J. Proteome analysis of chronically inflamed lungs in a mouse chronic asthma model. Int Arch Allergy Immunol. 2008;147(3):179-89. doi: 10.1159/000142040. Epub 2008 Jul 2. PMID 18594147
- [Background] Quesada Calvo F, Fillet M, Renaut J, Crahay C, Gueders M, Hacha J, Paulissen G, Foidart JM, Noel A, Rocks N, Leprince P, Cataldo D. Potential therapeutic target discovery by 2D-DIGE proteomic analysis in mouse models of asthma. J Proteome Res. 2011 Sep 2;10(9):4291-301. doi: 10.1021/pr200494n. Epub 2011 Aug 3. PMID 21751807
- [Background] Liao W, Goh FY, Betts RJ, Kemeny DM, Tam J, Bay BH, Wong WS. A novel anti-apoptotic role for apolipoprotein L2 in IFN-gamma-induced cytotoxicity in human bronchial epithelial cells. J Cell Physiol. 2011 Feb;226(2):397-406. doi: 10.1002/jcp.22345. PMID 20665705
- [Background] Fitzpatrick AM, Higgins M, Holguin F, Brown LA, Teague WG; National Institutes of Health/National Heart, Lung, and Blood Institute's Severe Asthma Research Program. The molecular phenotype of severe asthma in children. J Allergy Clin Immunol. 2010 Apr;125(4):851-857.e18. doi: 10.1016/j.jaci.2010.01.048. PMID 20371397